CLINICAL TRIAL: NCT01453296
Title: A Randomized, Double-blind, Placebo-controlled, Two-way Crossover 7-day Study to Investigate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Repeat Dose Inhaled GW642444 25 μg (Micrograms) in Children Aged 5-11 Years With Persistent Asthma.
Brief Title: Pharmacokinetics and Pharacodynamics of GW642444 in Paedetric Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 112776
Record Dates: First submitted 2011-09-01; First posted 2011-10-17 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Asthma; Tolerability; Safety; Pharmacokinetics; GW642444
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- COHORT 1 (RANDOMISATION AB or BA) (Active Comparator): 8-11 years old; Subjects will be assigned to receive GW642444 25μg or matching placebo (in a 1:1 ratio) in an AB or BA (A= GW64244, B= Placebo) sequence.
  Following randomisation (AB or BA) subjects will receive a single dose treatment, followed by 7 day washout period. This will then be followed by a repeat dose session of the same treatment (Day 8 and Day 14 in house, Days 9-13 at home).
  Each subject will then complete the same sequence for the alternative treatment in the second session. There will be a washout period of at least 7 days between the treatment periods.
  Interventions: Drug: GW642444; Drug: Placebo
- COHORT 2 (RANDOMISATION AB or BA) (Active Comparator): 5-7 years old. Subjects will be assigned to receive GW642444 25μg or matching placebo (in a 1:1 ratio) in an AB or BA (A= GW64244, B= Placebo) sequence.
  Following randomisation (AB or BA) subjects will receive a single dose treatment, followed by 7 day washout period. This will then be followed by a repeat dose session of the same treatment (Day 8 and Day 14 in house, Days 9-13 at home).
  Each subject will then complete the same sequence for the alternative treatment in the second session. There will be a washout period of at least 7 days between the treatment periods.
  Interventions: Drug: GW642444; Drug: Placebo

INTERVENTIONS:
Drug: GW642444 — GW642444 25 μg; Novel dry powder inhaler
Drug: Placebo — Matching placebo; Novel dry powder inhaler

SUMMARY:
This study will investigate the effect of dosing paedeatric asthmatic subjects with GW642444, an orally inhaled long-acting agonist of the β2-adrenoceptor.

DETAILED DESCRIPTION:
This study will investigate the effect of dosing with 25 μg GW642444, an orally inhaled long-acting agonist of the β2-adrenoceptor, in asthmatic subjects aged 5 to 11. GW642444 is currently under development as the long-acting beta-agonist component of a combination product containing an inhaled corticosteroid and a longacting beta-agonist.

Subjects will receive a single dose via a novel dry powder inhaler, then 7 days once-daily repeat dosing following a washout period. The study will be a randomized two-way crossover, with a placebo control. Approximately 26 subjects will be recruited to this study, with the aim that 20 will complete the study. Safety, tolerability, pharmacokinetics and glucose and potassium levels will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male and pre-menarchial female subjects aged 5-11 years on the last planned treatment day are eligible for this study. Pre-menarchial females are defined as any female who has yet to begin menses and is considered Tanner Stage 2 or less.
* Diagnosis of asthma at least 6 months prior to screening.
* Patients must be controlled on their existing asthma treatment at Screening as defined by a Childhood Asthma Control Test score of >19 and PEF (Peak Expiratory Flow) >75 % predicted.
* Subjects must be taking a stable regimen of fluticasone propionate (≤200 μg (micrograms) twice daily or equivalent) and short acting beta-agonist inhaler on an as-need basis for at least 4 weeks prior to screening.
* Apart from asthma, eczema and rhinitis, subjects should be healthy and suffer from no other significant medical conditions.
* Subjects must weigh at least 15 kg (kilograms).
* Subjects must demonstrate ability to accept and effectively use the GW642444 device using the demonstration kits provided to the site.
* The subject and parent or guardian are able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions. The parent or guardian must have the ability to read, write and record diary information collected throughout the study. The parent or guardian must also have the ability to manage study drug administration and PEF assessments.
* At least one parent or guardian has signed and dated the written informed consent prior to admission to the study. This will be accompanied by informed assent from the subject.

Exclusion Criteria:

* Subjects currently receiving (or have received within 4 weeks of screening) any of the following asthma therapies: theophyllines, long-acting inhaled beta-agonists, oral beta-agonist.
* Subjects who have changed their asthma medication within 4 weeks of screening.
* Clinical visual evidence of oral candidiasis at screening.
* Any clinically relevant abnormality identified on the screening medical assessment
* Any medical condition or circumstance making the subject unsuitable for participation in the study (e.g. history of life-threatening asthma)
* Asthma exacerbation requiring systemic corticosteroids (oral, intramuscular, intravenous) or Emergency Room attendance within 3 months or asthma exacerbation requiring hospitalization within 6 months prior to the screening visit.
* Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract which is not resolved within 4 weeks of the screening visit.
* Any adverse reaction including immediate or delayed hypersensitivity to any betaagonist therapy.
* Known or suspected sensitivity to the constituents of the novel dry powder inhaler (i.e., lactose or magnesium stearate), for example, history of severe milk protein allergy.
* The parent or guardian has history of psychiatric disease, intellectual deficiency, substance abuse, or other condition (e.g., inability to read, comprehend or write) which will limit the validity of consent to participate in this study.
* A subject will not be eligible for this study if he/she is an immediate family member of the participating Investigator, sub-Investigator, study coordinator, or employee of the participating Investigator.
* Children who are wards of the state or government.
* Evidence of clinically significant abnormality in the 12-lead ECG (electrocardiogram) at Screening

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - GSK Investigational Site, Cypress, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Medford, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 112776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112776 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into one of two cohorts based upon age; the younger cohort was enrolled after a review of the safety/pharmacokinetic data of at least six participants from the older cohort. Each participant was assigned to treatment randomly; assignment was not to be influenced by whether participants were in Cohort 1 or Cohort 2.
Pre-assignment Details: A Baseline assessment was carried out on Day 1 of the first treatment period. Participants were then randomized to one of the two possible treatment sequences (Vilanterol [VI] 25 micrograms [µg] followed by matching Placebo; matching placebo followed by VI 25 µg) in a 1:1 ratio in an AB or BA sequence.
Groups:
- Sequence 1: VI 25 µg Followed by Placebo: Participants received vilanterol (VI) 25 micrograms (µg) and matching placebo in Treatment Periods 1 and 2, respectively. Inhaled VI 25 µg and matching placebo were administered once daily in the morning (Day 1 to Day 14) via ae Dry Powder Inhaler. The washout period between the 14-day treatment periods was at least 7 days.
- Sequence 2: Placebo Followed by VI 25 µg: Participants received placebo and VI 25 µg in Treatment Periods 1 and 2, respectively. Inhaled VI 25 µg and matching placebo were administered once daily in the morning (Day 1 to Day 14) via a Dry Powder Inhaler. The washout period between the 14-day treatment periods was at least 7 days.
Period: Treatment Period 1
Arm/Group | Sequence 1: VI 25 µg Followed by Placebo | Sequence 2: Placebo Followed by VI 25 µg
Started | 14 | 14
Completed | 13 | 13
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Met Protocol-Defined Stopping Criteria | 1 | 0
Period: Washout Period
Arm/Group | Sequence 1: VI 25 µg Followed by Placebo | Sequence 2: Placebo Followed by VI 25 µg
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Sequence 1: VI 25 µg Followed by Placebo | Sequence 2: Placebo Followed by VI 25 µg
Started | 13 | 13
Completed | 11 | 13
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- VI 25 µg/Placebo or Placebo/VI 25 µg: Participants received either vilanterol (VI) 25 micrograms (µg) or matching placebo in the first of two 14-day treatment periods, followed by a repeat dose of the other therapy (the therapy not received in the first treatment period) in the second 14-day treatment period. Inhaled VI 25 µg or matching placebo was administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler. The washout period between the treatment periods was at least 7 days.
Arm/Group | VI 25 µg/Placebo or Placebo/VI 25 µg
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.0 (1.90)
Gender [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 5
  White - White/Caucasian/European Heritage | 22
  Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Any Serious Adverse Event (SAE) During the Treatment Period
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in deciding whether reporting is appropriate in other situations. Refer to the General AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From the start of study medication until Week 11 (Visit 8)/Early Withdrawal
Population: All Subjects Population: all participants who received at least one dose of study medication
Measure: Number; unit: Participants
Groups:
- Placebo: All participants who received matching placebo in one or both of the two 14-day treatment periods. Matching placebo was administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler. The washout period between the treatment periods was at least 7 days.
- VI 25 µg: All participants who received VI 25 µg in one or both of the 14-day treatment periods. Inhaled VI 25 µg was administered once daily in the morning (Day 1 to Day 14) via the Dry Powder Inhaler. The washout period between the treatment periods was at least 7 days.
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
Participants
  Any AE | 6 | 9
  Any SAE | 0 | 0

2. Primary Outcome: Basophil, Eosinophil, Lymphocyte, Monocyte, Total Neutrophil, Platelet, and White Blood Cell Count Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of basophils, eosinophils, lymphocytes, monocytes, total neutrophils, platelets, and white blood cell (WBC) count at Day 14 of the respective treatment period. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
10^9 cells per liter (GI/L)
  Basophils, n=24, 25 | 0.021 (0.0145) | 0.034 (0.0185)
  Eosinophils, n=24, 25 | 0.276 (0.3002) | 0.348 (0.3458)
  Lymphocytes, n=24, 25 | 2.404 (0.8652) | 2.419 (0.8729)
  Monocytes, n=24, 25 | 0.268 (0.1310) | 0.376 (0.1419)
  Total neutrophils, n=24, 25 | 3.354 (1.3054) | 3.127 (0.9625)
  Platelets, n=23, 25 | 280.7 (54.11) | 279.4 (54.71)
  WBCs, n=24, 25 | 6.32 (1.808) | 6.30 (1.640)

3. Primary Outcome: Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of hemoglobin and MCHC at Day 14 of the respective treatment period. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
Grams per liter (g/L)
  Hemoglobin, n=24, 25 | 133.0 (11.30) | 130.7 (11.22)
  MCHC, n=24, 25 | 337.1 (5.50) | 338.3 (11.60)

4. Primary Outcome: Reticulocyte and Red Blood Cell (RBC) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of reticulocytes and RBCs at Day 14 of the respective treatment period. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (TI/L)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
10^12 cells per liter (TI/L)
  Reticulocytes, n=24, 25 | 0.05010 (0.020696) | 0.05275 (0.024571)
  RBCs, n=24, 25 | 4.60 (0.374) | 4.47 (0.339)

5. Primary Outcome: Hematocrit Value at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of hematocrit at Day 14 of the respective treatment period. Hematocrit is a measure of the percentage of the volume of the whole blood that is composed of red blood cells, as determined by separation of red blood cells from the plasma (usually by centrifugation). Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: proportion of 1
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 24 | 25
proportion of 1 | 0.3948 (0.03430) | 0.3863 (0.02617)

6. Primary Outcome: Mean Corpuscle Volume (MCV) Value at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of MCV at Day 14 of the respective treatment period. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^15 femtoliters (fL) per cell
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 24 | 25
10^15 femtoliters (fL) per cell | 86.0 (4.08) | 86.6 (3.59)

7. Primary Outcome: Mean Corpuscle Hemoglobin (MCH) Value at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of MCH at Day 14 of the respective treatment period. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 picograms (pg) per cell
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 24 | 25
10^12 picograms (pg) per cell | 28.97 (1.337) | 29.29 (1.464)

8. Primary Outcome: Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), and Gamma Glutamyl Transferase (GGT) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of ALT, ALP, AST, and GGT at Day 14 of the respective treatment period. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: All Subjects Population, Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
International units per liter (IU/L)
  ALT, n=22, 25 | 13.9 (4.21) | 13.5 (3.56)
  ALP, n=22, 25 | 260.5 (109.65) | 273.4 (103.51)
  AST, n=22, 24 | 27.7 (6.11) | 25.5 (4.52)
  GGT, n=22, 25 | 14.1 (4.12) | 13.6 (3.51)

9. Primary Outcome: Albumin and Total Protein Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of albumin and total protein at Day 14 of the respective treatment period. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
Grams per liter
  Albumin, n=22, 25 | 42.8 (2.95) | 43.2 (1.96)
  Total protein, n=22, 25 | 67.9 (4.82) | 68.6 (3.16)

10. Primary Outcome: Calcium, Chloride, Carbon Dioxide (CO2) Content/Bicarbonate, Glucose, Potassium, Sodium, and Urea/Blood Urea Nitrogen (BUN) Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of calcium, chloride, carbon dioxide content/bicarbonate (CO2/BI), glucose, potassium, sodium, and urea/BUN at Day 14 of the respective treatment period. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
Millimoles per liter (mmol/L)
  Calcium, n=22, 24 | 2.327 (0.1357) | 2.359 (0.0666)
  Chloride, n=22, 25 | 105.5 (3.90) | 105.1 (2.01)
  CO2 content/bicarbonate, n=22, 24 | 17.6 (2.30) | 18.1 (1.98)
  Glucose, n=22, 25 | 4.95 (0.510) | 5.04 (0.513)
  Potassium, n=22, 24 | 4.30 (0.408) | 4.33 (0.242)
  Sodium, n=22, 25 | 137.7 (2.43) | 137.8 (2.12)
  Urea/BUN, n=22, 25 | 4.91 (1.368) | 4.48 (1.150)

11. Primary Outcome: Total Bilirubin, Direct Bilirubin, Creatinine, and Uric Acid Values at Day 14 of the Respective Treatment Period
Description: Blood samples were collected for the measurement of total bilirubin, direct bilirubin, creatinine, and uric acid at Day 14 of the respective treatment period. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
Micromoles per liter (µmol/L)
  Total bilirubin, n=22, 25 | 6.2 (2.22) | 5.8 (1.99)
  Direct bilirubin, n=22, 25 | 1.7 (0.94) | 1.2 (1.00)
  Creatinine, n=22, 25 | 39.45 (7.653) | 39.35 (6.731)
  Uric acid, n=22, 25 | 241.4 (69.51) | 245.6 (47.27)

12. Primary Outcome: Peak Expiratory Flow on Day 1, Day 8, and Day 14 of the Respective Treatment Period
Description: Peak Expiratory Flow (PEF) is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF is calculated as the maximum of three readings taken at each timepoint for each participant. Baseline is defined as the pre-dose measurement at Day 1 for the respective period. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg (n=28).
Time Frame: Day 1, Day 8, and Day 14 of the respective treatment period (up to Study Day 49)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different time points, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 28
liters/minute
  Day 1, Baseline, n=26, 28 | 230.6 (72.55) | 233.0 (68.55)
  Day 1, 20 minutes post-dose, n=26, 28 | 237.5 (69.65) | 245.6 (73.47)
  Day 8, Pre-dose, n=26, 28 | 232.1 (64.76) | 228.8 (64.42)
  Day 8, 20 minutes post-dose, n=25, 28 | 233.8 (220.0) | 240.7 (65.66)
  Day 14, Pre-dose, n=24, 26 | 240.3 (75.90) | 239.0 (72.02)
  Day 14, 20 minutes post-dose, n=24, 26 | 243.3 (75.18) | 248.1 (76.20)

13. Primary Outcome: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Day 1, Day 8, and Day 14 of the Respective Treatment Period
Description: SBP and DBP were measured at Day 1, Day 8, and Day 14 of the respective treatment period. PD=post-dose. Baseline is defined as the pre-dose measurement at Day 1 for the respective period. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg (n=28).
Time Frame: Day 1, Day 8, and Day 14 of the respective treatment period (up to Study Day 49)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 28
Millimeters of mercury (mmHg)
  Day 1 SBP, Baseline, n=26, 28 | 101.8 (6.59) | 102.9 (9.21)
  Day 1 SBP, 10 minutes PD, n=26, 28 | 100.7 (7.59) | 102.4 (7.69)
  Day 1 SBP, 30 minutes PD, n=26, 28 | 100.9 (9.35) | 103.5 (6.89)
  Day 1 SBP, 45 minutes PD, n=26, 28 | 100.9 (7.41) | 103.5 (7.05)
  Day 1 SBP, 74 minutes PD, n=26, 28 | 102.7 (7.95) | 104.4 (6.81)
  Day 1 SBP, 2 hours PD, n=26, 28 | 103.3 (8.16) | 104.8 (7.82)
  Day 8 SBP, Pre-dose, n=25, 28 | 99.6 (6.92) | 103.7 (8.64)
  Day 8 SBP, 30 minutes PD, n=25, 28 | 101.7 (7.29) | 102.9 (7.31)
  Day 8 SBP, 1 hour PD, n=25, 28 | 101.8 (8.38) | 103.6 (7.17)
  Day 14 SBP, Pre-dose, n=24, 26 | 101.5 (9.18) | 103.9 (6.15)
  Day 14 SBP, 10 minutes PD, n=24, 26 | 101.3 (9.98) | 103.7 (6.70)
  Day 14 SBP, 30 minutes PD, n=24, 26 | 103.9 (8.72) | 102.9 (8.91)
  Day 14 SBP, 45 minutes PD, n=24, 26 | 103.6 (7.95) | 103.4 (7.03)
  Day 14 SBP, 75 minues PD, n=24, 26 | 104.9 (8.33) | 103.9 (6.36)
  Day 14 SBP, 4 hours PD, n=24, 26 | 102.2 (7.80) | 106.0 (5.20)
  Day 14 SBP, 2 hours PD, n=24, 26 | 103.0 (6.68) | 102.9 (6.42)
  Day 14 SBP, 8 hours PD, n=24, 26 | 104.7 (8.92) | 104.7 (7.76)
  Day 1 DBP, Baseline, n=26, 28 | 62.0 (5.12) | 62.1 (6.38)
  Day 1 DBP, 10 minutes PD, n=26, 28 | 62.4 (7.16) | 63.5 (4.08)
  Day 1 DBP, 30 minutes PD, n=26, 28 | 62.4 (6.55) | 62.6 (4.29)
  Day 1 DBP, 45 minutes PD, n=26, 28 | 63.0 (7.93) | 63.3 (5.99)
  Day 1 DBP, 75 minutes PD, n=26, 28 | 63.3 (5.74) | 64.4 (7.91)
  Day 1 DBP, 2 hours PD, n=26, 28 | 63.0 (4.81) | 63.4 (5.49)
  Day 8 DBP, Pre-dose, n=25, 28 | 63.7 (8.17) | 62.8 (5.58)
  Day 8 DBP, 30 minutes PD, n=25, 28 | 62.3 (9.19) | 62.4 (7.26)
  Day 8 DBP, 1 hour PD, n=25, 28 | 63.2 (6.68) | 62.2 (7.90)
  Day 14 DBP, Pre-dose, n=24, 26 | 60.8 (5.70) | 63.8 (8.14)
  Day 14 DBP, 10 minutes PD, n=24, 26 | 60.9 (6.55) | 62.7 (7.07)
  Day 14 DBP, 30 minutes PD, n=24, 26 | 62.8 (3.83) | 63.7 (7.88)
  Day 14 DBP, 45 minutes PD, n=24, 26 | 61.9 (4.05) | 64.5 (4.68)
  Day 14 DBP, 75 minutes PD, n=23, 26 | 63.0 (5.12) | 63.6 (6.34)
  Day 14 DBP, 2 hours PD, n=23, 26 | 64.1 (7.33) | 63.3 (5.50)
  Day 14 DBP, 4 hours PD, n=23, 26 | 62.3 (8.56) | 63.9 (6.59)
  Day 14 DBP, 8 hours PD, n=23, 26 | 63.2 (4.78) | 63.3 (7.29)

14. Primary Outcome: Maximum Heart Rate at Day 1 and Day 14 of the Respective Treatment Period
Description: Heart rate (HR) was measured at Day 1 and Day 14 of the respective treatment period. hr=hour. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg (n=28).
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 28
Beats per minute
  Day 1 maximum HR (0-2 hr), n=26, 28 | 83.6 (1.44) | 86.1 (1.40)
  Day 14 maximum HR (0-2 hr), n=24, 26 | 84.3 (1.38) | 85.0 (1.35)
  Day 14 maximum HR (0-8 hr), n=24, 26 | 88.1 (1.45) | 88.6 (1.41)
Statistical Analysis 1: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-0.8 to 5.7] — Day 1 maximum HR (0-2 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo
Statistical Analysis 2: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-2.4 to 3.7] — Day 14 maximum HR (0-2 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-2.6 to 3.6] — Day 14 maximum HR (0-8 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo

15. Primary Outcome: Weighted Mean Heart Rate at Day 1 and Day 14 of the Respective Treatment Period
Description: Heart rate (HR) was measured at Day 1 and Day 14 of the respective treatment period. hr=hour. Weighted means were derived using the linear trapezoidal rule. Actual relative times were used for the calculation except where actual times were missing. If any actual times were missing, planned relative times were used for these observations. For 0-8 hr parameters, treatment, period, participant Baseline, and period Baseline were fitted as fixed effects, and participant was fitted as a random effect. For 0-2 hr parameters, treatment, period, day (1 and 14), participant Baseline, period Baseline, and treatment*day interaction were fitted as fixed effects, and participant was fitted as a random effect. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg (n=28).
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 28
Beats per minute
  Day 1 weighted HR (0-2 hr), n=26, 28 | 76.39 (1.311) | 79.20 (1.285)
  Day 14 weighted mean HR (0-2 hr), n=23, 26 | 76.11 (1.309) | 77.67 (1.264)
  Day 14 weighted mean HR (0-8 hr), n=23, 26 | 80.54 (1.458) | 80.65 (1.404)
Statistical Analysis 1: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-0.8 to 5.7] — Day 1 weighted HR (0-2 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo
Statistical Analysis 2: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-2.4 to 3.7] — Day 14 weighted HR (0-2 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-2.6 to 3.6] — Day 14 weighted HR (0-8 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo

16. Primary Outcome: Maximum QTcF at Day 1 and Day 14 of the Respective Treatment Period
Description: The electrocardiographic (ECG) parameter QT duration corrected using Fridericia's formula (QTcF) was measured at Day 1 and Day 14 of the respective treatment period. hr=hour. For 0-8 hr parameters, treatment, period, participant Baseline, and period Baseline were fitted as fixed effects, and participant was fitted as a random effect. For 0-2 hr parameters, treatment, period, day (1 and 14), participant Baseline, period Baseline, and treatment*day interaction were fitted as fixed effects, and participant was fitted as a random effect. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg (n=28).
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 28
milliseconds
  Day 1 maximum QTcF (0-2 hr), n=26, 28 | 405.6 (2.29) | 406.6 (2.22)
  Day 14 maximum QTcF (0-2 hr), n=24, 26 | 406.1 (2.06) | 407.7 (2.00)
  Day 14 maximum QTcF (0-8 hr), n=24, 26 | 407.8 (1.87) | 409.2 (1.82)
Statistical Analysis 1: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-4.5 to 6.6] — Day 1 maximum QTcF (0-2 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo
Statistical Analysis 2: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-3.2 to 6.3] — Day 14 maximum QTcF (0-2 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-3.0 to 5.7] — Day 14 maximum QTcF (0-8 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo

17. Secondary Outcome: AUC(0-t) and AUC(0-8) on Day 14 of the Respective Treatment Period
Description: Area under the concentration-time (AUC) curve from time zero (pre-dose) to the last time AUC(0-t) and from time zero to 8 hours AUC(0-8) of quantifiable concentration of VI on Day 14 of the respective treatment period was measured. Samples were collected at the following times: pre-dose; 10 minutes (min) and 30 min post-dose; and 1, 2, 4, 6, and 8 hours post-dose for participants who were >=20 kilograms and pre-dose; 10 min and 30 min post-dose; and 1, 2, and 4 hours post-dose for participants who were <=20 kilograms on Day 14 of the respective treatment period. Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the Pharmacokinetic Population.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: Pharmacokinetic (PK) Population: all participants in the All Subjects Population for whom a PK sample was obtained and analyzee. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: picograms*hour per milliliter (pg*hr/mL)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 0 | 25
picograms*hour per milliliter (pg*hr/mL)
  AUC(0-t), n=25 |  | 132.8 [96.0 to 183.8]
  AUC(0-8), n=19 |  | 181.7 [145.0 to 227.7]

18. Secondary Outcome: Cmax on Day 14 of the Respective Treatment Period
Description: Cmax is defined as the maximum observed concentration on Day 14 of the respective treatment period. Samples were collected at the following times: pre-dose; 10 minutes (min) and 30 min post-dose; and 1, 2, 4, 6, and 8 hours post-dose for participants who were >=20 kilograms and pre-dose; 10 min and 30 min post-dose; and 1, 2, and 4 hours post-dose for participants who were <=20 kilograms on Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: picograms per milliliter (pg/mL)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 0 | 25
picograms per milliliter (pg/mL) |  | 97.44 [64.83 to 146.45]

19. Secondary Outcome: Tmax, t1/2, and t at Day 14 of the Respective Treatment Period
Description: tmax is defined as the time to reach the observed maximum concentration, t1/2 is defined as the time required to reduce the plasma concentration to one half its initial value, and t is defined as the time of the last observed quantifiable concentration on Day 14 of the respective treatment period. Samples were collected at the following times: pre-dose; 10 minutes (min) and 30 min post-dose; and 1, 2, 4, 6, and 8 hours post-dose for participants who were >=20 kilograms and pre-dose; 10 min and 30 min post-dose; and 1, 2, and 4 hours post-dose for participants who were <=20 kilograms on Day 14 of the respective treatment period.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: PK Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the PK Population.
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 0 | 25
hours
  tmax, n=23 |  | 0.20 [0.00 to 1.00]
  t1/2, n=14 |  | 3.131 [1.06 to 6.32]
  t, n=23 |  | 6.00 [1.00 to 8.13]

20. Secondary Outcome: Blood Glucose and Potassium on Day 14 of the Respective Treatment Period
Description: Blood glucose and potassium values were measured on Day 14 of the respective treatment period. Samples were collected at the following times: pre-dose; 10 minutes (min) and 30 min post-dose; and 1, 2, 4, 6, and 8 hours post-dose for participants who were >=20 kilograms and pre-dose; 10 min and 30 min post-dose; and 1, 2, and 4 hours post-dose for participants who were <=20 kilograms on Day 14 of the respective treatment period. . Weighted means were derived using the linear trapezoidal rule. Actual relative times were used for the calculation except where actual times were missing. If any actual times were missing, planned relative times were used for these observations. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg. Treatment and period were fitted as fixed effects and participant was fitted as a random effect.
Time Frame: Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
Millimoles per liter (mmol/L)
  Maximum Glucose (0-2 hr), n=24, 26 | 5.55 (0.184) | 5.57 (0.182)
  Maximum Glucose (0-8 hr), n=24, 26 | 6.22 (0.187) | 6.03 (0.183)
  Weighted Mean Glucose (0-2 hr), n=21, 25 | 5.02 (0.114) | 5.06 (0.109)
  Weighted Mean Glucose (0-8 hr), n=19, 24 | 5.26 (0.108) | 5.21 (0.100)
  Minimum Potassium (0-2 hr), n=23, 26 | 4.05 (0.040) | 4.00 (0.038)
  Minimum Potassium (0-8 hr), n=24, 26 | 3.89 (0.060) | 3.87 (0.059)
  Weighted Mean Potassium (0-2 hr), n=19, 22 | 4.21 (0.049) | 4.23 (0.046)
  Weighted Mean Potassium (0-8 hr), n=17, 22 | 4.05 (0.052) | 4.11 (0.049)

21. Secondary Outcome: Average Oropharyngeal Cross-sectional Area on Day 1 and Day 14 of the Respective Treatment Period
Description: During the pharyngometry assessment, participants inhaled through a wavetube, which had a mouthpiece with the same dimensions as the mouthpiece on the dry powder inhaler used for the study. This technique was used to measure the size of the throat and mouth (oropharynx) in the form of pharyngograms. Pharyngometry data were recorded for each day (Day 1 and Day 14 of the respective treatment period) using the mean of four measurements (pharyngograms), and the average oropharyngeal cross-sectional area was calculated.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: All Subjects Population. Only those participants available at the specified time point were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: centimeters squared (cm^2)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
centimeters squared (cm^2)
  Day 1, n=15, 13 | 5.65 (1.834) | 4.42 (2.310)
  Day 14, n=14, 15 | 5.47 (1.661) | 5.16 (2.139)

22. Secondary Outcome: Distance of Assessment on Day 1 and Day 14 of the Respective Treatment Period
Description: During the pharyngometry assessment, participants inhaled through a wavetube, which had a mouthpiece with the same dimensions as the mouthpiece on the dry powder inhaler used for this study. This technique was used to measure the size of the throat and mouth (oropharynx) in the form of pharyngograms. Distance of assessment is defined as the distance (length measured in centimeters [cm]) estimated to be from the lips to the larynx. Pharyngometry data were recorded for each day (Days 1 and 14 of the respective treatment period) using the mean of four measurements (pharyngograms), and the average oropharyngeal cross-sectional area was calculated.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
centimeters (cm)
  Day 1, n=15, 13 | 18.40 (1.502) | 18.26 (1.824)
  Day 14, n=14, 15 | 18.46 (1.395) | 18.41 (1.276)

23. Secondary Outcome: Oropharyngeal Volume on Day 1 and Day 14 of the Respective Treatment Period
Description: During the pharyngometry assessment, participants inhaled through a wavetube, which had a mouthpiece with the same dimensions as the mouthpiece on the dry powder inhaler used for this study. This technique was used to measure the size of the throat and mouth (oropharynx) in the form of pharyngograms. Oropharyngeal volume is defined as the volume (centimeters cubed [cm^3]) of the mouth and throat estimated to be from the lips to the larynx. Pharyngometry data were recorded for each day (Days 1 and 14 of the respective treatment period) using the mean of four measurements (pharyngograms), and the average oropharyngeal cross-sectional area was calculated.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
cm^3
  Day 1, n=15, 13 | 102.33 (32.451) | 78.60 (39.296)
  Day 14, n=14, 15 | 102.26 (36.322) | 93.35 (37.190)

24. Secondary Outcome: Average Flow Rate and Peak Inspiratory Flow Rate (PIFR) on Day 1 and Day 14 of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Average flow rate is defined as the average inspiratory flow rate (Liters [L]/min) across the inhalation profile when inhaling across the resistance of the inhaler. PIFR is defined as the Peak Inspiratory Flow Rate (L/min) of the inhalation profile when inhaling across the resistance of the inhaler.The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was used for each day (Days 1 and 14 of the respective treatment period), and the average flow rate and PIFR were determined. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Liters per minute (L/min)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
Liters per minute (L/min)
  Day 1, Average flow rate, n=23, 25 | 38.84 (9.440) | 42.23 (10.952)
  Day 14, Average flow rate, n=23, 25 | 40.45 (10.538) | 42.08 (10.191)
  Day 1, PIFR, n=23, 25 | 58.27 (14.258) | 61.41 (16.513)
  Day 14, PIFR, n=23, 25 | 60.93 (14.901) | 61.79 (15.348)

25. Secondary Outcome: Inhalation Time on Day 1 and Day 14 of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Inhalation time is defined as the duration of the inhalation(s) when inhaling across the resistance of the inhaler. The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was used for each day (Days 1 and 14 of the respective treatment period), and the inhalation time was determined. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Seconds (sec)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
Seconds (sec)
  Day 1, n=23, 25 | 1.45 (0.604) | 1.36 (0.551)
  Day 14, n=23, 25 | 1.35 (0.528) | 1.34 (0.476)

26. Secondary Outcome: Inhaled Volume on Day 1 and Day 14 of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Inhaled volume is defined as the volume of air (Liters) inhaled during the inhalation across the resistance of the inhaler.
  The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was used for each day (Days 1 and 14 of the respective treatment period), and the inhalaled volume was determined. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
Liters
  Day 1, n=23, 25 | 0.93 (0.433) | 0.92 (0.343)
  Day 14, n=23, 25 | 0.90 (0.426) | 0.95 (0.417)

27. Secondary Outcome: Peak Pressure Drop on Day 1 and Day 14 of the Respective Treatment Period
Description: During the inhalation profile assessment, participants inhaled through a mouthpiece from a device with a similar resistance to the dry powder inhaler used for this study. Peak pressure drop is defined as the maximum pressure drop (kilopascal [kPa]) achieved during inhalation across the resistance of the inhaler. The pressure drop during the inhalation was measured, and the inhalation profiles (pressure drop versus time profile) of the participants were obtained. The mean of the two inhalation profile measurements was calculated for each day (Days 1 and 14 of the respective treatment period), and used for subsequent modeling and prediction of dose emission attributes. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Kilopascal (kpa)
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 27
Kilopascal (kpa)
  Day 1, n=23, 25 | 2.97 (1.275) | 3.33 (1.632)
  Day 14, n=23, 25 | 3.23 (1.479) | 3.33 (1.350)

28. Secondary Outcome: Total Emitted Dose (TED) on Day 1 and Day 14 of the Respective Treatment Period
Description: The total emitted dose (TED) is defined as the mass (micrograms) of the nominal dose that passes beyond the throat. The recorded inhalation profiles of the participants and the mouth-throat (oropharyngeal) models of the sizes that approximated to pharyngometry measurements of the participants were used in conjunction with the electronic Lung (eLung) for in vitro assessment. The eLung is a breathing simulator that replicates the selected inhalation profile with an active inhaler placed at the lips end of the selected ororpharyngeal model. After the dose is emitted from the inhaler, the analysis and assay of throat deposition and material passing beyond the throat was used to derive the nominal, minimum, and maximum predicted total emitted dose.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: All Subjects Population. Only those participants available at the specified time point were analyzed. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg.
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 0 | 25
micrograms
  Nominal TED |  | 20.28 (0.177)
  Minimum TED |  | 20.24 (0.188)
  Maximum TED |  | 20.31 (0.173)

29. Secondary Outcome: Ex-throat Dose (ETD) and ETD <2 Microns on Day 1 and Day 14 of the Respective Treatment Period
Description: The ex-throat dose (ETD) and the "nominal ETD" is the mass (micrograms) of active investigational material that passes beyond the throat, nominal being the mean.The recorded inhalation profiles of the participants and the mouth-throat (oropharyngeal) models of the sizes that approximated to pharyngometry measurements of the participants were used in conjunction with the electronic Lung (eLung) for in vitro assessment. The eLung is a breathing simulator that replicates the selected inhalation profile with an active inhaler placed at the lips end of the selected ororpharyngeal model. After the dose is emitted from the inhaler, the analysis and assay of throat deposition and material passing beyond the throat was used to derive the nominal, minimum, and maximum predicted ETD and ETD <2 microns.
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: All Subjects Population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 0 | 15
micrograms
  Nominal ETD |  | 9.00 (0.697)
  Minimum ETD |  | 8.94 (0.652)
  Maximum ETD |  | 9.06 (0.747)
  ETD <2 microns |  | 4.19 (1.079)
  Minimum ETD <2 microns |  | 4.10 (1.011)
  Maximum ETD <2 microns |  | 4.29 (1.157)

30. Primary Outcome: Weighted Mean QTcF at Day 1 and Day 14 of the Respective Treatment Period
Description: The electrocardiographic (ECG) parameter QT duration corrected using Fridericia's formula (QTcF) was measured at Day 1 and Day 14 of the respective treatment period. hr=hour. Actual relative times were used for the calculation except where actual times were missing. If any actual times were missing, planned relative times were used for these observations. For 0-8 hr parameters, treatment, period, participant Baseline, and period Baseline were fitted as fixed effects, and participant was fitted as a random effect. For 0-2 hr parameters, treatment, period, day (1 and 14), participant Baseline, period Baseline, and treatment*day interaction were fitted as fixed effects, and participant was fitted as a random effect. Subject 2308 received VI 25 µg in both treatment periods, and contributed twice to the summary of VI 25 µg (n=28).
Time Frame: Day 1 and Day 14 of the respective treatment period (up to Study Day 49)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Placebo | VI 25 µg
Number analyzed (Participants) | 26 | 28
milliseconds
  Day 1 weighted mean QTcF (0-2 hr), n=26, 28 | 394.21 (2.007) | 396.22 (1.960)
  Day 14 weighted mean QTcF (0-2 hr), n=23, 26 | 395.09 (2.122) | 398.03 (2.024)
  Day 14 weighted mean QTcF (0-8 hr), n=23, 26 | 393.43 (1.867) | 396.62 (1.793)
Statistical Analysis 1: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.01, 95% CI 2-sided [-2.59 to 6.61] — Day 1 weighted QTcF (0-2 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo
Statistical Analysis 2: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 2.94, 95% CI 2-sided [-1.93 to 7.81] — Day 14 weighted QTcF (0-2 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo
Statistical Analysis 3: Comparison: Placebo vs VI 25 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.19, 95% CI 2-sided [-0.70 to 7.08] — Day 14 weighted QTcF (0-8 hr). The estimated value represents the treatment difference: VI 25 µg minus placebo

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and non-serious AEs were collected in members of the All Subjects Population, comprised of all participants who received at least one dose of study medication.
Arm/Group | Placebo | VI 25 µg
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 6/26 | 9/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | VI 25 µg (N=27)
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Otitis media (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Pyrexia (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.